CLINICAL TRIAL: NCT00094770
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of the Addition of MK0431 Compared With Sulfonylurea Therapy in Patients With Type 2 Diabetes With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: An Investigational Drug Study in Patients With Type 2 Diabetes Mellitus (0431-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-024; MK0431-024; 2004_049
Record Dates: First submitted 2004-10-22; First posted 2004-10-25 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin 100 mg (Experimental): Sitagliptin 100 mg oral tablets of sitagliptin once daily.
  Interventions: Drug: sitagliptin (MK0431)
- Glipizide (Active Comparator): Glipizide 1 tablet (5 mg) per day. Patients could then up-titrated to a total daily dose of 4 tablets twice daily (20mg/day) based on their glycemic control.
  Interventions: Drug: Comparator: glipizide

INTERVENTIONS:
Drug: sitagliptin (MK0431) — Sitagliptin 100 mg oral tablets of sitagliptin once daily.
  Other Names: MK0431
  Arms: Sitagliptin 100 mg
Drug: Comparator: glipizide — Glipizide 1 tablet (5 mg) per day. Patients could then up-titrated to a total daily dose of 4 tablets twice daily (20mg/day) based on their glycemic control.
  Other Names: Glipizide
  Arms: Glipizide

SUMMARY:
The purpose of this investigational study is to determine the safety and effectiveness of an investigational drug in patients with type 2 diabetes mellitus (a specific type of diabetes).

DETAILED DESCRIPTION:
The duration of treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age and not older than 78 with type 2 diabetes mellitus

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Nauck MA, Meininger G, Sheng D, Terranella L, Stein PP; Sitagliptin Study 024 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor, sitagliptin, compared with the sulfonylurea, glipizide, in patients with type 2 diabetes inadequately controlled on metformin alone: a randomized, double-blind, non-inferiority trial. Diabetes Obes Metab. 2007 Mar;9(2):194-205. doi: 10.1111/j.1463-1326.2006.00704.x. PMID 17300595
- [Derived] Ommen ES, Xu L, O'Neill EA, Goldstein BJ, Kaufman KD, Engel SS. Comparison of treatment with sitagliptin or sulfonylurea in patients with type 2 diabetes mellitus and mild renal impairment: a post hoc analysis of clinical trials. Diabetes Ther. 2015 Mar;6(1):29-40. doi: 10.1007/s13300-015-0098-y. Epub 2015 Jan 30. PMID 25633134
- [Derived] Seck TL, Engel SS, Williams-Herman DE, Sisk CM, Golm GT, Wang H, Kaufman KD, Goldstein BJ. Sitagliptin more effectively achieves a composite endpoint for A1C reduction, lack of hypoglycemia and no body weight gain compared with glipizide. Diabetes Res Clin Pract. 2011 Jul;93(1):e15-7. doi: 10.1016/j.diabres.2011.03.006. Epub 2011 Apr 8. PMID 21477878
- [Derived] Seck T, Nauck M, Sheng D, Sunga S, Davies MJ, Stein PP, Kaufman KD, Amatruda JM; Sitagliptin Study 024 Group. Safety and efficacy of treatment with sitagliptin or glipizide in patients with type 2 diabetes inadequately controlled on metformin: a 2-year study. Int J Clin Pract. 2010 Apr;64(5):562-76. doi: 10.1111/j.1742-1241.2010.02353.x. PMID 20456211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 26-Oct-2004; Last Patient Last Visit: 17-May-2007; 173 medical clinics worldwide.
Pre-assignment Details: Participants 18-78 years of age with type 2 diabetes mellitus (T2DM) and inadequate glycemic control (Hemoglobin A1c >6.5% and < 10%) on metformin at a dose of >1500mg/day.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily.
- Glipizide: The Glipizide group includes data from patients randomized to receive treatment with glipizide initiated at a dose of 1 tablet (5 mg) per day. Patients could then up-titrated to a total daily dose of 4 tablets twice daily (20mg/day) based on their glycemic control.
Period: Year 1 ( Week 0 to Week 52)
Arm/Group | Sitagliptin 100 mg | Glipizide
Started | 588 | 584
Completed | 386 (4 Participants who Completed Week 52, Did NOT Enter second year) | 412 (11 Participants who Completed Week 52, Did NOT Enter second year)
Not Completed | 202 | 172
Not completed — Adverse Event | 25 | 26
Not completed — Lack of Efficacy | 86 | 58
Not completed — Lost to Follow-up | 19 | 10
Not completed — Protocol Violation | 10 | 10
Not completed — Protocol Specified Discontinuation | 19 | 25
Not completed — Patient Moved | 6 | 2
Not completed — Withdrawal by Subject | 25 | 28
Not completed — Site Terminated | 2 | 2
Not completed — Other | 10 | 11
Period: Year 2 (Week 0 to Week 104)
Arm/Group | Sitagliptin 100 mg | Glipizide
Started | 588 | 584
Completed | 255 | 264
Not Completed | 333 | 320
Not completed — Adverse Event | 35 | 36
Not completed — Lack of Efficacy | 180 | 162
Not completed — Lost to Follow-up | 25 | 15
Not completed — Protocol Violation | 13 | 12
Not completed — Protocol Specified Discontinuation | 29 | 30
Not completed — Patient Moved | 6 | 2
Not completed — Withdrawal by Subject | 28 | 38
Not completed — Site Terminated | 2 | 2
Not completed — Other | 15 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Glipizide | Total
Number analyzed (Participants) | 588 | 584 | 1172
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.3) | 56.6 (9.8) | 56.7 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 226 | 478
  Male | 336 | 358 | 694
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 50 | 49 | 99
  Black | 41 | 35 | 76
  Hispanic | 43 | 46 | 89
  White | 432 | 434 | 866
  Other | 22 | 20 | 42
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.7 (0.9) | 7.6 (0.9) | 7.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 52
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 52 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and Week 52
Population: The per protocol population required that a participant had measurements both at baseline and at Week 52, and did not have any major protocol violations (e.g. drug compliance < 75%, addition of prohibited antihyperglycemic agent, incorrect double-blind study medication). No missing data were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 382 | 411
Percent | -0.67 [-0.75 to -0.59] | -0.67 [-0.75 to -0.59]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 104
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 104 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and Week 104
Population: The per protocol population required that a participant had measurements both at baseline and at Week 104, and did not have any major protocol violations (e.g. drug compliance < 75%, addition of prohibited antihyperglycemic agent, incorrect double-blind study medication). No missing data were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 248 | 256
Percent | -0.54 [-0.64 to -0.45] | -0.51 [-0.60 to -0.42]

3. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: Change from baseline at Week 52 is defined as Week 52 minus Week 0.
Time Frame: Baseline and Week 52
Population: The All-Patient-as-Treated (APaT) population required that a participant received at least 1 dose of double-blind study therapy. No missing data were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 389 | 416
Kilograms | -1.5 [-2.0 to -0.9] | 1.1 [0.5 to 1.6]

4. Secondary Outcome: Change From Baseline in Body Weight at Week 104
Description: Change from baseline at Week 104 is defined as Week 104 minus Week 0.
Time Frame: Baseline and Week 104
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 253 | 261
Kilograms | -1.6 [-2.3 to -1.0] | 0.7 [0.0 to 1.3]

5. Secondary Outcome: Hypoglycemic Events at Week 52
Description: Number of participants who reported 1 or more episodes of the adverse experience (AEs) of hypoglycemia.
Time Frame: Baseline to Week 52
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  Participants with one or more Hypoglycemic AEs | 29 | 187
  Total number of Hypoglycemic episodes | 50 | 657
  Participants with no Hypoglycemic AEs | 559 | 397

6. Secondary Outcome: Hypoglycemic Events at Week 104
Description: Number of participants who reported 1 or more episodes of the adverse experience of hypoglycemia.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  Participants with one or more Hypoglycemic AEs | 31 | 199
  Total number of Hypoglycemic episodes | 57 | 805
  Participants with no Hypoglycemic AEs | 557 | 385

7. Secondary Outcome: Number of Participants With Clinical Adverse Experiences (CAEs) at Week 104
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  With CAES | 452 | 480
  Without CAES | 136 | 104

8. Secondary Outcome: Number of Participants With Serious CAEs at Week 104
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  With serious CAEs | 64 | 73
  Without serious CAEs | 524 | 511

9. Secondary Outcome: Number of Participants With Drug-related CAEs at Week 104
Description: Participants with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  With drug related CAEs | 97 | 193
  Without drug related CAEs | 491 | 391

10. Secondary Outcome: Number of Participants With Laboratory Adverse Experiences (LAEs) at Week 104
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  With LAEs | 85 | 74
  Without LAEs | 503 | 510

11. Secondary Outcome: Number of Participants With Serious LAEs at Week 104
Description: Serious LAEs are any LAEs occurring at any dose that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants
  With serious LAEs | 0 | 0
  Without serious LAEs | 588 | 584

12. Secondary Outcome: Number of Participants With Drug-related LAEs at Week 104
Description: Participants with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) LAEs.
Time Frame: Baseline to Week 104
Population: All randomized participants who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Glipizide
Number analyzed (Participants) | 588 | 584
Participants | 18 | 21

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg | Glipizide
Serious Adverse Events (participants affected / at risk) | 64/588 | 73/584
Other Adverse Events (participants affected / at risk) | 318/588 | 374/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=588) | Glipizide (N=584)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Angina Pectoris (Cardiac disorders) | 1 | 3
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Hypertensive Heart Disease (Cardiac disorders) | 1 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 2 | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Macular Hole (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal Polyp (Gastrointestinal disorders) | 1 | 0
Splenic Artery Aneurysm (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Oedema Peripheral (General disorders) | 1 | 0
Polyserositis (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden Cardiac Death (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Abdominal Wall Abscess (Infections and infestations) | 0 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Dengue Fever (Infections and infestations) | 0 | 1
Diabetic Foot Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 1
Medical Device Complication (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 2
Multiple Injuries (Injury, poisoning and procedural complications) | 2 | 0
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Intraocular Pressure Increased (Investigations) | 0 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Astrocytoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Carcinoid Tumour Of The Small Bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Neoplasm Malignant Non-Resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Mass (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Extremity Necrosis (Vascular disorders) | 0 | 1
Iliac Artery Stenosis (Vascular disorders) | 1 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0
Venous Insufficiency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=588) | Glipizide (N=584)
Diarrhoea (Gastrointestinal disorders) | 42 | 40
Bronchitis (Infections and infestations) | 40 | 37
Influenza (Infections and infestations) | 32 | 37
Nasopharyngitis (Infections and infestations) | 71 | 61
Upper Respiratory Tract Infection (Infections and infestations) | 73 | 79
Urinary Tract Infection (Infections and infestations) | 44 | 25
Hypoglycaemia (Metabolism and nutrition disorders) | 31 | 199
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 32
Back Pain (Musculoskeletal and connective tissue disorders) | 35 | 32
Headache (Nervous system disorders) | 33 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 32
Hypertension (Vascular disorders) | 29 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.